CLINICAL TRIAL: NCT05432999
Title: Effect of Extracorporeal Shockwave Therapy on Spasticity in Chronic SCI: A Pilot Study
Brief Title: Extracorporeal Shockwave Therapy for Spasticity in People With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nathan Hogaboom, PhD, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1178-22
Record Dates: First submitted 2022-06-23; First posted 2022-06-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Spasticity, Muscle; Spastic Paraplegia; Spastic Quadriplegia; Spastic Tetraplegia; Paraplegia; Tetraplegia
Keywords: shockwave; extracorporeal shockwave therapy; spinal cord injury; spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity; Paraplegia; Quadriplegia | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial with sham control
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): This group will receive a focused extracorporeal shockwave therapy treatment (three applications over three weeks), applied to the spastic medial gastrocnemius.
  Interventions: Device: Extracorporeal Shockwave Therapy
- Control (Sham Comparator): This group will go through the same procedures as the intervention group, but the shockwave device will not touch their skin and thus they will receive no therapeutic effect.
  Interventions: Device: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — Shockwaves are high pressure sound waves that interact with tissues to elicit a biological response. The shockwave probe will be placed on the skin with ultrasound gel and the muscle will be stimulated for a few minutes.
  Other Names: Storz Medical DUOLITH SD1 Ultra modular system

SUMMARY:
People with spinal cord injury (SCI) experience a host of secondary complications that can impact their quality of life and functional independence. One of the more prevalent complications is spasticity, which occurs in response to spinal cord damage and the resulting disruption of motor pathways. Common symptoms include spasms and stiffness, and can occur more than once per hour in many people with SCI. Spasticity can have a negative impact over many quality of life domains, including loss of functional independence, activity limitations, and even employment. Its impact on health domains is also pronounced, with many people who have spasticity reporting mood disorders, depression, pain, sleep disturbances, and contractures. Spasticity can interfere with post-injury rehabilitation and lead to hospitalization. There are many treatments for spasticity in this population. However, many do not have long-term efficacy, and, if they do, they are often pharmacological in nature and carry side effects that could limit function or affect health. The goal of this pilot, randomized-controlled study is to investigate the potential efficacy and safety of a non-invasive treatment with a low side effect profile, extracorporeal shockwave therapy (ESWT). ESWT has shown some benefits in people with post-stroke spasticity with no long term side effects. Thirty individuals with chronic, traumatic SCI will be recruited. Fifteen will be provided with ESWT while the other fifteen will be given a sham treatment. Clinical and self-report measures of spasticity and its impact on quality of life will be collected, as well as quantitative ultrasound measures of muscle architecture and stiffness. The ultimate goal of this pilot project is to collect the data necessary to apply for a larger randomized-controlled trial. Conducting a larger trial will allow for a more powerful estimation of safety and efficacy of ESWT as a treatment for spasticity in people with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Have a non-progressive traumatic SCI (complete or incomplete) with residual neurological deficits that occurred greater than 1 year prior to their enrollment.
3. MAS score of 2 or greater in the gastrocnemius of the treated limb.
4. Can be treated with shockwaves. Contraindications include current or recent (within the past 3 months) infection at the site of treatment and severe coagulopathies (e.g. hemophilia).164
5. No change in antispasmodic medications within the past three months or intended changes over the course of the trial.
6. Participant is able and willing to comply with the protocol.

Exclusion Criteria:

1. History of surgical procedures of the lower extremity.
2. Ankle contracture.
3. Sever, inflammatory arthritic diseases.
4. Thrombosis.
5. Anticoagulant medications.
6. Pregnancy.
7. Cancer.
8. Recent history of local injection of botulinum toxin within 6 months, or phenol/alcohol with 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Ashworth Scale scores | 4 weeks
  The Modified Ashworth Scale (MAS) is a physical exam maneuver used frequently both clinically and for research purposes to assess the increase in velocity-dependent muscle tone after neurologic disorders. We will be focusing on the MAS score of the ankle plantar flexors. This measure is included in the NINDS list of CDE recommendations for SCI. Specifically, it evaluates the resistance to passive stretch of the ankle joint through full range of motion.

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale scores | 8 weeks
  The Modified Ashworth Scale (MAS) is a physical exam maneuver used frequently both clinically and for research purposes to assess the increase in velocity-dependent muscle tone after neurologic disorders. We will be focusing on the MAS score of the ankle plantar flexors. This measure is included in the NINDS list of CDE recommendations for SCI. Specifically, it evaluates the resistance to passive stretch of the ankle joint through full range of motion.
Change in Modified Tardieu Scale | 4 weeks
  The Modified Tardieu Scale (MTS) was developed as a more accurate method to measure spasticity by assessing muscle tone at different velocities. Since its development, it has gone through multiple modifications. The MTS is also included in the NINDS CDE recommendations as a measure of spasticity in people with SCI. The MTS includes two measurements, quality and angle of muscle reaction.
Change in Modified Tardieu Scale | 8 weeks
  The Modified Tardieu Scale (MTS) was developed as a more accurate method to measure spasticity by assessing muscle tone at different velocities. Since its development, it has gone through multiple modifications. The MTS is also included in the NINDS CDE recommendations as a measure of spasticity in people with SCI. The MTS includes two measurements, quality and angle of muscle reaction.
Change in Modified Penn Spasticity Frequency Scale | 4 weeks
  The Modified Penn Spasticity Frequency Scale (mPSFS) is a self-report scale with two components, which is meant to provide a more complete understanding of an individual's spasticity status. The first component is comprised of a five-point scale, which assesses spasm frequency between 0 ("no spasms") and 4 ("spontaneous spasms occurring more than 10 times per hour"). The second component includes a three-point scale, which assesses spasm severity between 1 ("mild") and 3 ("severe"); this component is not answered if the individual reports no spasms in part one.
Change in Modified Penn Spasticity Frequency Scale | 8 weeks
  The Modified Penn Spasticity Frequency Scale (mPSFS) is a self-report scale with two components, which is meant to provide a more complete understanding of an individual's spasticity status. The first component is comprised of a five-point scale, which assesses spasm frequency between 0 ("no spasms") and 4 ("spontaneous spasms occurring more than 10 times per hour"). The second component includes a three-point scale, which assesses spasm severity between 1 ("mild") and 3 ("severe"); this component is not answered if the individual reports no spasms in part one.
Change in Modified Patient-Reported Impact of Spasticity Measure | 4 weeks
  The Modified Patient-Reported Impact of Spasticity Measure (mPRISM) is a self-reported instrument with 37 items that assesses the impact of spasticity on health-related quality of life. It is separated into physical, psychological, and social subdomains, making is possible to investigate how spasticity impacts different aspects of quality of life. Each item is rated using a scale of 0 ("never") to 3 ("often to very often").
Change in Modified Patient-Reported Impact of Spasticity Measure | 8 weeks
  The Modified Patient-Reported Impact of Spasticity Measure (mPRISM) is a self-reported instrument with 37 items that assesses the impact of spasticity on health-related quality of life. It is separated into physical, psychological, and social subdomains, making is possible to investigate how spasticity impacts different aspects of quality of life. Each item is rated using a scale of 0 ("never") to 3 ("often to very often").
Participant Global Impression of Change | 4 weeks
  The Participant Global Impression of Change (PGIC, also referred to as the original Guy-Farrar/PGIC scale) is used to measure global treatment effect. It asks the participant to rate, using a 7-point scale (anchored by "very much worse" and "very much improved"), his or her overall impression following treatment as compared to before the treatment. This scale is particularly useful as it provides an indication of clinically important improvement. Although it was designed for and has commonly been used in pain trials, it has been used to assess efficacy of spasticity treatments in people with SCI.
Participant Global Impression of Change | 8 weeks
  The Participant Global Impression of Change (PGIC, also referred to as the original Guy-Farrar/PGIC scale) is used to measure global treatment effect. It asks the participant to rate, using a 7-point scale (anchored by "very much worse" and "very much improved"), his or her overall impression following treatment as compared to before the treatment. This scale is particularly useful as it provides an indication of clinically important improvement. Although it was designed for and has commonly been used in pain trials, it has been used to assess efficacy of spasticity treatments in people with SCI.
Medial gastrocnemius muscle echogenicity | 4 weeks
  Average "brightness" of the medial gastrocnemius muscle, measured using quantitative ultrasound techniques.
Medial gastrocnemius muscle echogenicity | 8 weeks
  Average "brightness" of the medial gastrocnemius muscle, measured using quantitative ultrasound techniques.
Medial gastrocnemius muscle elasticity | 4 weeks
  Average elasticity of the medial gastrocnemius muscle, measured using shear wave elastography.
Medial gastrocnemius muscle elasticity | 8 weeks
  Average elasticity of the medial gastrocnemius muscle, measured using shear wave elastography.
Medial gastrocnemius muscle fiber length | 4 weeks
  Fiber length of the medial gastrocnemius muscle, measured quantitatively using ultrasound.
Medial gastrocnemius muscle fiber length | 8 weeks
  Fiber length of the medial gastrocnemius muscle, measured quantitatively using ultrasound.
Medial gastrocnemius muscle thickness | 4 weeks
  Thickness of the medial gastrocnemius muscle, measured quantitatively using ultrasound.
Medial gastrocnemius muscle thickness | 8 weeks
  Thickness of the medial gastrocnemius muscle, measured quantitatively using ultrasound.
Medial gastrocnemius muscle pennation angle | 4 weeks
  Pennation angle of the medial gastrocnemius muscle, measured quantitatively using ultrasound.
Medial gastrocnemius muscle pennation angle | 8 weeks
  Pennation angle of the medial gastrocnemius muscle, measured quantitatively using ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No